CLINICAL TRIAL: NCT01710306
Title: Web and Shared Decision Making for Reserve/National Guard Women's PTSD Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CRE 12-039
Record Dates: First submitted 2012-09-21; First posted 2012-10-19 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: PTSD
Keywords: Women; Veterans; PTSD; Access to Care; Shared Decision Making
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outreach (No Intervention): To evaluate and test differences in VA mental health care engagement for those who screen positive for PTSD by randomly assigned route: existing OEF/OIF/OND outreach. VA mental health care engagement is defined as participation in any of the following: PTSD psychotherapy, cognitive processing therapy, or prolonged exposure therapy.
- Nurse Care Manager (NCM) (Experimental): To evaluate and test differences in VA mental health care engagement for those who screen positive for PTSD by randomly assigned route: Study concierge nurse case manager (NCM). VA mental health care engagement is defined as participation in any of the following: PTSD psychotherapy, cognitive processing therapy, or prolonged exposure therapy.
  Interventions: Behavioral: Nurse Care Manager (NCM)

INTERVENTIONS:
Behavioral: Nurse Care Manager (NCM) — Nurse care manager interventions with telephone implemented shared decision making protocol compared to outreach as usual OEF/OIF/OND outreach.
  Arms: Nurse Care Manager (NCM)

SUMMARY:
Women and Reserve/National (RNG) Veterans are among the fastest growing groups of new VA users. While PTSD is prevalent in this group, most women don't access or complete needed treatment. This study will investigate Operation enduring/Iraqi Freedom and New Dawn (OEF/OIF/OND) RNG female war Veterans' perceptions, preferences, barriers and facilitators to accessing VA mental health (MH) and evidence-based PTSD psychotherapy. This information will be used to revise an existing web-based screen that educates participants about their unique post-deployment MH conditions. This web-interface will then be used to randomly assign women who screen positive for PTSD to either 1) a concierge nurse case manager who uses shared decision-making to engage Veterans in EBP or 2) usual outreach to determine what engagement approach women prefer. The investigators' findings will provide VA leaders with key information to understand and improve access to RNG PTSD treatment.

DETAILED DESCRIPTION:
Women and OEF/OIF/OND Reserve/National Guard (RNG) war Veterans are among the fastest growing groups of new VA users. Although PTSD is highly prevalent in this group of Veterans, most choose not to seek care for a variety of reasons. Facilitating access to mental health (MH) services for RNG OEF/OIF/OND female Veterans with post-traumatic stress disorder (PTSD) is challenging and requires new approaches to outreach. Such approaches are urgently needed to mediate the severity of post-deployment MH conditions, alleviate concerns over MH diagnoses, and interrupt the cycle of chronicity found in many with PTSD. This gap between need for and use of VA PTSD services suggests that further research is needed to understand specific barriers to VA mental health (MH) care and VA PTSD evidence-based psychotherapy (EBP). A web-based interface tailored to consumer needs has the potential to promote active engagement by Veterans in their health care. Considering that OEF/OIF combat Veterans enrolled in VA care report a preference to seek readjustment services or information over the internet, such an approach may have important advantages for engaging this group. Furthermore, evidence indicates that when patients are educated about their physical health conditions and treatment alternatives, shared decision-making results in increased treatment participation, better adherence to treatment recommendations, and better health outcomes. Although highly promising, web-based and shared-decision making approaches to facilitating VA MH treatment utilization are in need of further study.

In Phase 1 of the project, the investigators will use qualitative methods to assess VA enrolled PTSD positive OEF/OIF/OND RNG female war Veterans' perceptions, preferences and barriers and facilitators to accessing VA MH services and evidence based psychotherapy (EBP) for PTSD. This information will be used to refine the investigators' existing web-based interface to better address these issues. Satisfaction with the revised interface will then be assessed. Phase 2 will focus on comparing the efficacy of two approaches to promoting VHA initiation. Participants who screen positive for PTSD on the web interface will be randomly assigned to: 1) Study concierge nurse case manager (NCM) facilitated shared decision making to assist with VA MH evaluation and treatment; or 2) existing outreach (current standard of care). Follow-up assessments will be conducted at 6 and 12 months to determine whether and where participants sought MH care (from both VA and non-VA resources).

This study will provide valuable insights about this population's perceptions of VA MH services and of PTSD EBP, as well as their evolving use of VA and other community resources to address PTSD and other post-deployment MH needs. Furthermore, it will provide important information regarding the efficacy of relatively inexpensive and resource-sparing interventions that can be readily implemented within existing and emerging (e.g., Patient Alight Care Teams [PACT]) models of VA care delivery. While the proposed web interface and shared decision-making intervention are currently directed at RNG women Veterans post-deployment, there are clear implications for expansion to other populations and health/MH concerns, as well. Findings have important policy implications for several operational partners heavily invested in the improved access and delivery of evidence-based mental health care for Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* R/NG servicewomen who have returned from deployment in service of and/or to Iraq/Afghanistan within the last 60 months.

Exclusion Criteria:

* Any disability that would impair individuals ability to provide consent and participate in the interview.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne G. Sadler, PhD RN, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Outreach: To evaluate and test differences in VA initiation and use for those who screen positive for PTSD by randomly assigned route: existing OEF/OIF/OND outreach. That is, VA usual outreach by existing OEF/OIF/OND transition patient advocates.
- Study Concierge Nurse Case Manager (NCM): To evaluate and test differences in VA initiation (did they seek VA care - new or return visit) and for participants who screen positive for PTSD they will be randomly assigned to either: 1)Study nurse case manager (NCM) or outreach as usual..
  NCM: Nurse care manager interventions will consist of telephone delivered shared decision protocols with participants compared to OEF/OIF/OND outreach as usual.
Period: Overall Study
Arm/Group | Outreach | Study Concierge Nurse Case Manager (NCM)
Started | 86 | 85
Completed | 68 | 55
Not Completed | 18 | 30

BASELINE CHARACTERISTICS:
Groups:
- Outreach: To evaluate and test differences in VA mental health care engagement for those who screen positive for PTSD by randomly assigned route: existing OEF/OIF/OND outreach. VA mental health care engagement is defined as participation in any of the following: PTSD psychotherapy, cognitive processing therapy, or prolonged exposure therapy. That is, VA existing outreach by existing OEF/OIF/OND transition patient advocates.
- Study Concierge Nurse Case Manager (NCM): To evaluate and test differences in VA mental health care engagement for those who screen positive for PTSD by randomly assigned route: Study concierge nurse case manager (NCM). VA mental health care engagement is defined as participation in any of the following: PTSD psychotherapy, cognitive processing therapy, or prolonged exposure therapy.
- Total: Total of all reporting groups
Arm/Group | Outreach | Study Concierge Nurse Case Manager (NCM) | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.3) | 36.5 (9.7) | 36.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 85 | 171
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 15 | 25
  White | 57 | 48 | 105
  More than one race | 11 | 18 | 29
  Unknown or Not Reported | 8 | 4 | 12
Mental Health Care Engagement [Count of Participants; unit: Participants] | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With VA Mental Health Care Engagement
Description: VA mental health care engagement is defined as participation in any of the following: PTSD psychotherapy, cognitive processing therapy, or prolonged exposure therapy. To be identified in VA electronic medical record
Time Frame: Outcome measures are assessed at baseline interview and within 6 and 12 months following this semi-structured telephone interview .
Measure: Count of Participants; unit: Participants
Groups:
- Nurse Care Manger Intervention Arm: To evaluate and test differences in VA mental health care engagement for those who screen positive for PTSD by randomly assigned route: Study concierge nurse case manager (NCM). VA mental health care engagement is defined as participation in any of the following: PTSD psychotherapy, cognitive processing therapy, or prolonged exposure therapy.
Arm/Group | Outreach | Nurse Care Manger Intervention Arm
Number analyzed (Participants) | 86 | 85
Participants
  Engaged in Mental Health Care | 40 | 30
  Did Not Engage in Mental Health Care | 28 | 28
  Did Not Complete Participation | 18 | 27
Statistical Analysis 1: Comparison: Outreach vs Nurse Care Manger Intervention Arm; Test type: Superiority; p = 0.1996, Chi-squared

2. Secondary Outcome: Patient Activation Measure
Description: The Patient Activation Measure (PAM) administered on line to RCT participants yields a patient activation score allowing comparison of patient activation with other populations/studies The PAM-13 item measures patient knowledge, skill, and confidence for medical self-management. It is scored on a scale from 0-100. These scores result in four levels of patient activation that range from 1 to 4 with 1 being the lowest level of patient activation for taking action and 4 the highest level of activation. Specifically: 1=believing the patient role is important. 2=having confidence/knowledge necessary to take action. 3=actually taking action to maintain/improve one's health. 4=maintaining health actions, even under stress. The percentage of participants in each arm who had a PAM score that indicated a level of activation/taking action (levels 3 and 4) will be identified.
Time Frame: Outcome measure was assessed at baseline data collection
Population: Percentage of participants listed below are those in each arm who had a PAM score indicating a level of taking action (levels 3 and 4).
Measure: Count of Participants; unit: Participants
Arm/Group | Outreach | Nurse Care Manager (NCM)
Number analyzed (Participants) | 86 | 85
Participants | 50 | 53

ADVERSE EVENTS:
Time Frame: All study phases, years 1-4.
Arm/Group | Outreach | Study Concierge Nurse Case Manager (NCM)
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/85
Other Adverse Events (participants affected / at risk) | 0/86 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT01710306/Prot_SAP_000.pdf